CLINICAL TRIAL: NCT03766594
Title: Effect of Preconceptional Sildenafil Citrate Treatment in Women With Early Unexplained Recurrent Pregnancy Loss: a Randomized Controlled Trial
Brief Title: Sildenafil Citrate in Early Unexplained Recurrent Pregnancy Loss
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Yakout Mohamed, Resident of O&G, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SURPL
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Miscarriage, Recurrent
MeSH Terms: conditions — Abortion, Habitual | interventions — Sildenafil Citrate; Folic Acid

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups: Group (A) folic acid and sildenafil citrate and Group (B) folic acid and placebo.
  Folic acid (0.5 mg) will be started 3 months before conception in the two groups. Sildenafil citrate (dose: 25 mg; oral tablets, 4 times/day) or placebo will be started preconception for 24 days
Who Masked: Participant, Care Provider
Masking Description: Patients are randomized to receive either folic acid and sildenafil citrate or folic acid and placebo. Placebo tablets were same size and appearance of the sildenafil citrate tablets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sildenafil group (Active Comparator): Includes 45 women who received Sildenafil citrate (Respatio(R) 25mg tablets four times daily for 24 days preconceptionally starting first day of previous period) and folic acid (Folic acid(R) 0.5mg tablets once daily for 3 months preconceptionally).
  Interventions: Drug: Sildenafil Citrate; Drug: Folic Acid
- Control group (Active Comparator): Includes 45 women who received placebo oral tablets (apparently identical to Respatio(R) 25mg tablets, four times daily for 24 days preconceptionally starting first day of previous period) and folic acid (Folic acid(R) 0.5mg tablets once daily for 3 months preconceptionally).
  Interventions: Drug: Folic Acid; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Sildenafil Citrate — Respatio(R) 25mg tablets four times daily for 24 days preconceptionally starting first day of previous period
  Arms: Sildenafil group
Drug: Folic Acid — Folic acid(R) 0.5mg tablets once daily for 3 months preconceptionally
Drug: Placebo Oral Tablet — Placebo tablet apparently identical to Respatio(R) 25mg tablets, taken four times daily for 24 days preconceptionally starting first day of previous period
  Arms: Control group

SUMMARY:
Recurrent unexplained spontaneous miscarriage (RSM) is defined as three consecutive pregnancy loss prior to 20 weeks from the last menstrual period. 1% to 2% of women experience RSM. Treatment of URSM is a challenging issue. The currently available lines of treatment according to simplicity of use, reliability and degree of invasiveness include corticosteroids, sildenafil citrate, aspirin, heparin and immunoglobulins (besides good antenatal care), but up to now there are no prospective randomized studies, powerful enough, to determine a significant difference between these therapeutic protocols, with any of the above mentioned pharmacological agents.

Sildenafil Citrate (Viagra®), a vasodilator, is also described as an anti-inflammatory agent. While improving uterine blood flow in the proliferative phase, NO may have detrimental effects at the level of the endometrium during the implantation window. The NO- mediated release of cytokines such as tumour necrosis factor- from activated natural killer cells has been implicated as a cause of implantation failure.

Based on these observations, this study attempts was made to study uterine arteries and sub-endometrial blood flow during the luteal phase in normal fertile women and in patients with Unexplained recurrent miscarriage

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-35 years.
* BMI (20-30)
* History of three or more successive unexplained recurrent miscarriage.
* Normal uterine cavity by hystrography or hysteroscopy.
* No luteal phase defects by progesterone > 10 ng.
* Normal thyroid function (TSH, T3, T4)
* Normal lupus anticoagulant measured by activated partial throbmoplastine time (32-43 seconds).
* Normal anticardolipin (IgG < 20 gpl and IgM < 15 MPL measured by ELISA).
* Normal anti thyroid antibodies.
* Normal glucouse tolerance test.
* Normal parental karyotyping.

Exclusion Criteria:

* Age<20 or>35 year
* BMI<20 or>30
* Systemic diseases that might affect pregnancy such as diabetes or thyroid disorders or hypertension.
* History of consanguinity.
* Family history of chromosomal abnormalities (e.g. trisomy 21, trisomy 13, Turner's disease …etc.).
* History of autoimmune diseases, eg: systemic lupus.
* Congenital anomaly in uterine cavity as bicornate or septate uterus.
* Luteal phase defect and corpus luteum insufficiency.
* Uterine masses as fibroid or polyps.
* Patient with patuoles os.
* patient with antiphosphlipid syndrome.
* Cigarette smoking and alcohol.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Miscarriage rate | 24 gestational weeks
  number of spontaneous/missed miscarriages among the participants in both groups

SECONDARY OUTCOMES:
Uterine artery resistance index | At 24 gestational weeks
  Uterine artery resistance index assessed by uterine artery Doppler study in ongoing pregnancies of both groups
Uterine artery pulsatility index | At 24 gestational weeks
  Uterine artery pulsatility index assessed by uterine artery Doppler study in ongoing pregnancies of both groups

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Yakout, MBBCh, Principal Investigator — M Yakout
Locations (1):
- Ain SHams Maternity Hospital, Cairo, Abbaseya, Egypt